CLINICAL TRIAL: NCT00739284
Title: A Prospective Comparison Between Ureteral Stent and Nephrostomy Tube for an Urgent Drainage of Obstructed Kidney
Acronym: JJVsPCN08
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Dr. Shay Golan, Rabin medical center, Urology department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JJVsPCN08
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Kidney Disease
Keywords: preferred; procedure; drainage; obstructed; kidney; stone
MeSH Terms: conditions — Kidney Diseases; Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: nephrostomy tube and ureteral stent

SUMMARY:
Kidney obstruction might be caused by a stone in the urinary tract. In case of accompanying fever or renal failure, an urgent drainage might be needed. This can be done either by placing an ureteral stent or a nephrotomy tube. Only limited number of studies examined the question which of the two is preferred. A debate exist regarding the effectiveness of each procedure to improve symptoms, renal function and treating an infection. Our goal is to resolve this debate and to state whether one way is preferred on the other.

ELIGIBILITY:
Inclusion Criteria: Patient suffering from obstructed kidney by a stone and at least one of these situations:

1. fever (above 38c)
2. A rise in creatine to above 1.5
3. Pain resistent to multiple analgetic treatments

Exclusion Criteria:

* Patients with medical condition that prevent the use of one of the procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin medical center, Petah Tikva, Israel